CLINICAL TRIAL: NCT00148161
Title: Evoked and Induced Auditory Cortical Activity During Speech Perception and Speech Production in Stuttering
Brief Title: Activity of the Auditory Cortex During Speech Perception and Speech Production in Stuttering
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Other Study IDs: phonpaed001
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2006-09

CONDITIONS: Stuttering
Keywords: Magnetoencephalography; Auditory cortex; Stuttering; Non stuttering
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The goal of the study is to examine the cortical activity during speech perception and speech production in idiopathic stutterers compared to fluent speakers. Therefore, the noninvasive method of magnetoencephalography (MEG) is used. A better understanding for the complexity of speech perception and its pathology should be developed.

Fundamental properties of stuttering are repetitions, prolongations, and blocks. In most cases stuttering emerges between 2 and 5 years of age. The auditory feedback should become less important during development, as soon as information about mispronounced words does not occur anymore. During speech development this control function should be adopted by other systems. In stutterers the dominance of the acoustic control should remain.

Brain imaging studies with positron emission tomography (PET) or magnetic resonance imaging (MRI) show defects in the network of motor system, in the lateralization of speech areas, and functions of the auditory cortex. Magnetoencephalographic studies describe a similar variety as cause of stuttering. There may be defects in the auditory feedback, a modification of the lateralization of speech areas, or an alteration of co-action of motor planning and auditory system.

The benefit of magnetoencephalography is a very good temporal resolution in the range of milliseconds combined with good spatial resolution. Therefore, it is well suited to examine the dynamics of cortical processing during stuttering. In this study evoked components of the auditory systems related to complex sounds, vocals, consonant-vocal combinations, and single words are analyzed. Differences of these components in the auditory cortices of stutterers and fluent speakers are hypothesized as well in temporal structure as in localization and lateralization.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with idiopathic stuttering (for the group of stutterers)
* Fluently speaking subjects (for the control group)
* Right handed
* Normal hearing

Exclusion Criteria:

* Neurological diseases
* Psychiatric diseases
* Medication with neurological effective drugs
* Implants with magnetic impact

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette G Dinnesen, Prof. Dr., Study Director — Department of Phoniatrics and Pediatric Audiology, University Hospital Münster; Arne Knief, Dr., Principal Investigator — Department of Phoniatrics and Pediatric Audiology, University Hospital Münster
Locations (2):
- Germany (2):
  - Institute for Biomagnetism and Biosignalanalysis, Münster
  - Department of Phoniatrics and Pediatric Audiology, University Hospital Münster, Münster

REFERENCES:
- See also: Homepage of the Institute for Biomagnetism and Biosignalanalysis — http://biomag.uni-muenster.de